CLINICAL TRIAL: NCT04112693
Title: Assessment of the Neuro-glio-epithelial Unit (NGEU) in Biopsies Taken During Peroral Endoscopic Myotomy (POEM) for Achalasia: a Feasibility and Safety Study.
Acronym: Achalaglie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Rennes University Hospital (Other); University Hospital, Angers (Other Government); LA ROCHE SUR YON HOSPITAL (Unknown); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC19_0051
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Achalasia
Keywords: Achalasia; peroral endoscopic myotomy; neuro-glio-epithelial unit
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal biopsies during POEM (Experimental): In total, 14 biopsies are performed with a pediatric biopsy forceps belonging to the study center: 3 biopsies at 3-6 cm above cardia, contralaterally from POEM, of which 2 are placed in nitrogen and 1 in formol for histopathological analysis; 3 biopsies at the cardia, contralaterally from POEM, of which 2 are placed in nitrogen and 1 in formol for histopathological analysis; 4 biopsies of the muscularis propria (exposed during POEM) at 3-6 cm above cardia, of which 3 are placed in nitrogen and 1 in formol for histopathological analysis; 4 biopsies of the muscularis propria at the cardia, of which 3 are placed in nitrogen and 1 in formol for histopathological analysis; The biopsies for histopathological analysis will be analyzed in Full Field Optical Coherence Tomographie (FFOCT) before that. The FFOCT analysis take place for patient inclued after than 10 nov 2020.
  The biopsies are taken by the gastroenterologist who performs the POEM assisted by an endoscopy-specialized nurse.
  Interventions: Procedure: Esophageal biopsies during Peroral Endoscopic Myotomy (POEM)

INTERVENTIONS:
Procedure: Esophageal biopsies during Peroral Endoscopic Myotomy (POEM) — In total, 14 biopsies are performed with a pediatric biopsy forceps belonging to the study center: 3 biopsies at 3-6 cm above cardia, contralaterally from POEM, of which 2 are placed in nitrogen and 1 in formol for histopathological analysis; 3 biopsies at the cardia, contralaterally from POEM, of which 2 are placed in nitrogen and 1 in formol for histopathological analysis; 4 biopsies of the muscularis propria (exposed during POEM) at 3-6 cm above cardia, of which 3 are placed in nitrogen and 1 in formol for histopathological analysis; 4 biopsies of the muscularis propria at the cardia, of which 3 are placed in nitrogen and 1 in formol for histopathological analysis; The biopsies intended for histopathological analysis will be analyzed in FFOCT before histopathological analysis. The FFOCT analysis take place for the patient inclued after than 10 november 2020.
  The biopsies are taken by the gastroenterologist who performs the POEM and is assisted by an endoscopy-specialized nurse.

SUMMARY:
Achalasia is a primary esophageal motility disorder characterized on high-resolution manometry (HRM) studies by 100% failed peristalsis and elevated integrated relaxation pressure of the lower esophageal sphincter. It is further divided into 3 sub-types according to the Chicago classification v3.01. The pathophysiology of achalasia is poorly understood; however, the NGEU is increasingly recognized as playing a key role in the development of this disorder. Similarly, the esophageal muscle tissue is probably involved, but its sampling remained challenging until the recent advent of the POEM procedure. Indeed, it is now possible, easy and safe to take biopsies of the muscle tissue during POEM. Therefore, POEM not only represents an innovative and effective treatment for achalasia, but also an opportunity to better understand its underlying pathophysiological mechanisms. Currently available treatments for achalasia (pneumatic dilation (PD), Heller's myotomy (HM), botox injections, POEM) are "palliative" procedures that do not restore normal contractile function of the esophagus, but a better understanding of the pathophysiological mechanisms underlying this disorder could potentially help developing curative, or even preventative treatments.

To date, muscle tissue sampled during a POEM has only been characterized qualitatively (normal, atrophic, hypertrophic) with no assessment of the enteric nervous system. Moreover, there has been no studies of the mucosal or NGEU anomalies on biopsies taken during a minimally invasive procedure for achalasia such as a POEM.

This study aims to evaluate the feasibility of the assessment of NGEU and esophageal muscle tissue in biopsies taken during a POEM for achalasia. It also aims to determine whether specific biomarkers within the NGEU and muscle tissue can predict a better therapeutic response to a POEM. The goal is to include 30 patients within 12 months. Given that approximately 100 new cases of achalasia are diagnosed each year at the included centers, and that about 50% of treatment-naive patients are offered and accept to undergo a POEM, recruitment should be completed relatively rapidly. All POEMs will be performed at the CHU de Nantes by a single endoscopist who has already performed more than 100 procedures. Other than the complications related to the POEM itself, the addition of 14 esophageal biopsies required for our study is a very low-risk intervention. Biopsy sampling extends the length of the procedure by only 4-5 minutes and has not been associated with an increased risk of complications in a previous study.

Patients will be evaluated at five time points: preinclusion visit (up to four months before the POEM), inclusion visit (day of the POEM), post-POEM phone calls (3-6, 9-12, 22-26 months after POEM). During the preinclusion visit, relevant information regarding inclusion/exclusion criteria, consent, HRM and pH impedance results, past medical history, and pregnancy status (if applicable) will be gathered. At each time point, current medical history, Eckhardt score2 and pH impedance results (if available) will be documented. The patient will also answer the quality of life (SF36)3 and nutritional status questionnaires and will undergo blood sampling for albumin and prealbumin levels. Additionally, on the day of the POEM, there will be another blood sampling for complete blood count, PT, APTT, serum electrolytes and CRP level. Finally, at each post-POEM phone calls, the occurrence of adverse events will be reported.

Our primary hypothesis is that the analysis of mucosal and muscle tissue biopsies taken safely during a POEM will allow better characterization of transcriptomic and molecular remodeling of the mucosa (especially the NGEU) and the muscularis propria in achalasia. We also hypothesize that these anomalies could eventually serve as treatment targets and as a way of better stratifying patients according to achalasia type and treatment (in our case, POEM) response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years and above;
* Woman of child-bearing age, if using active (oral contraceptive pill, intrauterine device, contraceptive implant) and/or mechanical (condom, diaphragm) contraceptive method;
* Treatment-naive (no pneumatic dilation, botox injection, Heller's myotomy) patient with HRM-diagnosed achalasia in whom POEM is indicated;
* Thorough oral and written information about the protocol has been provided and patient's consent to participate in the study has been obtained;
* The patient is insured under the French social security system.

Exclusion Criteria:

* Active anticoagulant treatment or coagulation disorder
* Past history of achalasia treatment (pneumatic dilation, botox injection, Heller's myotomy)
* Pregnancy or breastfeeding
* Patient under trusteeship, guardianship, placed under judicial protection, and/or unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of the assessment of the NGEU and esophageal muscle tissue in biopsies taken during a POEM for achalasia. | Day 0
  Percentage of patients in whom the molecular and transcriptomic analyses of the NGEU and esophageal muscle tissue are possible

OTHER OUTCOMES:
Feasibility of the assessment of Full Field Optical Coherence Tomographie analysis of the mucosa and esophageal muscle | Day 0
  percentage of patients for whom FFOCT analysis of the mucosa and esophageal muscle is possible.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ARCHAMBEAUD, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes UH, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJ, Pandolfino JE; International High Resolution Manometry Working Group. The Chicago Classification of esophageal motility disorders, v3.0. Neurogastroenterol Motil. 2015 Feb;27(2):160-74. doi: 10.1111/nmo.12477. Epub 2014 Dec 3. PMID 25469569
- [Result] Eckardt VF, Aignherr C, Bernhard G. Predictors of outcome in patients with achalasia treated by pneumatic dilation. Gastroenterology. 1992 Dec;103(6):1732-8. doi: 10.1016/0016-5085(92)91428-7. PMID 1451966
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914